CLINICAL TRIAL: NCT02854709
Title: Effects of Sleep Extension on Glucose Metabolism in Chronically Sleep Deprived Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Sirimon Reutrakul, Associate Professor, Ramathibodi Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 065912
Record Dates: First submitted 2016-07-30; First posted 2016-08-03 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Sleep Extension; Glucose Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Continue with habitual sleep duration
- Intervention (Experimental): Sleep extension
  Interventions: Behavioral: Sleep extension

INTERVENTIONS:
Behavioral: Sleep extension — Sleep extension by 1 hour for 2 weeks
  Arms: Intervention

SUMMARY:
This is a randomized cross over study of the effect of 2-week sleep extension in chronically sleep deprived non-diabetic individuals on glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* self-reported sleep duration =<6 hours/night during the week with a desire to sleep at least 7 hours/night

Exclusion Criteria:

* shift workers,
* diabetes history,
* drugs affecting sleep or glucose metabolism,
* insomnia symptoms,
* high risk for sleep apnea,
* smoking or excess alcohol use

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism | 2 weeks
  Glucose and insulin values from 75 gram OGTT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Bangkok, Thailand